CLINICAL TRIAL: NCT04471441
Title: Multi-center, Open-label, Randomized Controlled Phase 4 Study to Evaluate the Efficacy and Safety of CertiroBell® Compared With Mycophenolate Mofetil in Primary Living Donor Liver Transplant Recipients.
Brief Title: Efficacy and Safety of Everolimus Versus Mycophenolate Mofetil in Liver Transplant Recipients.
Acronym: MONTBLANC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B95-02LT1903
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Liver Transplant
Keywords: Everolimus; CertiroBell; Mycophenolate mofetil
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CertiroBell Tablet (Experimental): De novo liver transplant recipients will be randomized after liver transplant operation.
  Interventions: Drug: Everolimus Tab.
- Mycophenolate mofetil Tablet/Capsule (Active Comparator): De novo liver transplant recipients will be randomized after liver transplant operation.
  Interventions: Drug: Mycophenolate mofetil Tab./Cap.

INTERVENTIONS:
Drug: Everolimus Tab. — After first dose 1mg BID(total 2mg daily PO), check the blood concentration of everolimus at each visit and adjust the dose to acheive the blood concentration maintaining at 3~8ng/mL.
  Other Names: CertiroBell Tab.
  Arms: CertiroBell Tablet
Drug: Mycophenolate mofetil Tab./Cap. — Up to 1.5g BID(total 3g daily), PO
  Arms: Mycophenolate mofetil Tablet/Capsule

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of CertiroBell® tablet compared with mycophenolate mofetil in primary living donor liver transplant recipients.

DETAILED DESCRIPTION:
This study is multi-center, open-label, randomized controlled phase 4 study to evaluate the efficacy and safety of certirobell® tablet compared with mycophenolate mofetil in primary living donor liver transplant recipients.

On the first visit the patients scheduled to be operated liver transplant in 35 days will be conducted screening. Patients who meet the criteria of this clinical trial will be randomized to CertiroBell or mycophenolate mofetil on the second visit. Each group will take CertiroBell or mycophenolate mofetil and will conduct scheduled tests with 5 additional visits.

ELIGIBILITY:
* Inclusion Criteria:

[Time of screening]

* Patients who have transplanted in primary living donor liver in 35 days or who plan to be transplanted in primary living donor liver.
* Over 20 years old(male or female)
* Agreement with written informed consent

[Time of randomization] - Patients who have transplanted liver within 4 weeks(25 days to 35 days)

* Exclusion Criteria

[Time of screening]

* Patients who have transplanted non-liver organs or have plan to be transplanted non-liver organs.
* Patients with bioartificial liver (cell system)
* Patients who diagnosed with malignant tumor within 5 years [however, who have recovered from skin cancer (squamous cell/basal cell carcinoma) or thyroid cancer, hepatocellular carcinoma without main vessel invasion or extrahepatic metastasis can be enrolled]
* Patients with severe systemic infection
* Women who are pregnant or breast feeding or not agree to the proper use of contraception during the trial
* Participated in other trial within 4 weeks
* In investigator's judgement

[Time of randomization]

* Patients with acute rejection who have been clinically treated after liver transplantation.
* Patients with complication related to the hepatic artery such as hepatic artery thrombosis at the time of randomization.
* At screening

  * WBC <1,500/mm^3 or PLT <30,000/mm^3 or over 3 times upper than normal range of liver function tests(T-bilirubin, AST, ALT) levels
  * Protein/Creatinine ratio(urine test) > 1 or eGFR by MDRD< 30mL/min/1.73m^2 or Total cholesterol > 350mg/dL or triglycerides > 500mg/dL
* Patients taking HCV(hepatitis C virus) Therapeutic Drugs
* Patients who had plasmapheresis within 1 week.
* Patents who had a record of taking mTOR inhibitor before.
* In investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-09-13 (Estimated); Study Completion 2022-11-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite efficacy failure | until 24 weeks after taking medicine
  composite efficacy failure include biopsy-confirmed acute rejection, graft loss, death, or follow-up failure

SECONDARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection | until 24weeks and 48weeks after taking medicine
  acute rejection confirmed by result of biopsy(over 4 points of RAI score)
The pathological results and time of occurrence and method of treatment, result of the treatment of acute rejection confirmed by biopsy(over 4 points of RAI score) | until 24weeks and 48weeks after taking medicine
  details of acute rejection confirmed by result of biopsy(over 4 points of RAI score)
Incidence of composite efficacy failure | until 48weeks after taking medicine
  composite efficacy failure include biopsy-confirmed acute rejection, graft loss, death, or follow-up failure
Survival rate of patients | until 24weeks and 48weeks after taking medicine
  Survival rate of patients
Survival rate of transplanted organ | until 24weeks and 48weeks after taking medicine
  Survival rate of transplanted organ
Incidence and recurrence rates of liver cancer | until 24weeks and 48weeks after taking medicine
  Incidence and recurrence rates of liver cancer
Incidence and recurrence rates of HCV infection | until 24weeks and 48weeks after taking medicine
  Incidence and recurrence rates of HCV infection
Incidence of CMV infection | until 24weeks and 48weeks after taking medicine
  Incidence of CMV infection
variation of Serum creatinine, eGFR(estimated glomerular filtration rate) compared to the baseline | at 24 weeks and 48weeks
  eGFR using MDRD(Modification of Diet in Renal Disease) method

CONTACTS AND LOCATIONS:
Overall Officials: Soon Il Kim, M.D., Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea